CLINICAL TRIAL: NCT06496815
Title: The Efficacy and Safety of Donafenib Combined With Immunotherapy and Local Therapy for Unresectable Hepatocellular Carcinoma That Has Failed in Previous Therapy
Brief Title: Donafenib Combined With Immunotherapy and Local Therapy for Unresectable Hepatocellular Carcinoma That Has Failed in Previous Therapy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zhiyong Huang, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: uHCC-Dona-TJ01
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Donafenib
MeSH Terms: interventions — donafenib; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donafenib combined with or without immunotherapy and local therapy for uHCC (Experimental): The patients who had previously received a targeted drug in combination with or without immunotherapy, local therapy (transhepatic arterial embolization chemotherapy (TACE), hepatic arterial infusion chemotherapy (HAIC)) and had not received donafenib, and the previous treatment has progressed. The specific experimental protocol was to replace the original targeted drug with donafenib (0.2g bid), while continuing immunotherapy and local therapy as previous (if have).
  Interventions: Drug: Donafenib; Procedure: transhepatic arterial embolization chemotherapy or hepatic arterial infusion chemotherapy; Drug: PD-1,PD-L1

INTERVENTIONS:
Drug: Donafenib — Donafenib will be taken orally twice a day, 0.2g each time.
Procedure: transhepatic arterial embolization chemotherapy or hepatic arterial infusion chemotherapy — Eligible subjects will receive transhepatic arterial embolization chemotherapy or hepatic arterial infusion chemotherapy as previous (if have).
Drug: PD-1,PD-L1 — PD-1/PD-L1 will be used as previous (if have).

SUMMARY:
The goal of this clinical trial is to learn if donafenib combined with or without immunotherapy and local therapy works to treat unresectable hepatocellular carcinoma that has failed in previous therapy.

It will also learn about the safety of donafenib combined with immunotherapy and local therapy.

The main questions it aims to answer are:

The Objective Response Rate (mRecist） and Progression-Free Survival of the participants treated by donafenib combined with immunotherapy and local therapy.

The disease control rate and overall survival of the participants treated by donafenib combined with immunotherapy and local therapy.

The safety of donafenib combined with immunotherapy and local therapy in the participants.

Participants will:

Replace the original targeted drug with donafenib (0.2g bid), while continuing immunotherapy and local therapy as previous therapy (if have).

The observation period was 1 year.

DETAILED DESCRIPTION:
This is a single-arm, prospective clinical study. 32 patients who had previously received a targeted drug in combination with or without immunotherapy, local therapy (transhepatic arterial embolization chemotherapy (TACE), hepatic arterial infusion chemotherapy (HAIC)) and had not received donafenib will be enrolled. The specific experimental protocol was to replace the original targeted drug with donafenib (0.2g bid), while continuing immunotherapy and local therapy as previous therapy(if have).The observation period was 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study, sign the informed consent form, and be aged between 18 and 70 years old.
2. Have at least one measurable lesion.
3. Clinically and pathologically diagnosed with hepatocellular carcinoma and not suitable for surgical resection.
4. Child-Pugh liver function classification: Class A/Class B.
5. Have previously received targeted therapy (excluding donafenib) in combination or not in combination with immunotherapy, locoregional therapy (transarterial chemoembolization (TACE), hepatic arterial infusion chemotherapy (HAIC)), and have clear tumor progression assessed by two clinicians using the RECIST criteria.
6. If infected with hepatitis B virus (HBV), such as positive for HBsAg, HBV-DNA must be tested, and HBV-DNA must be less than 500 IU/mL; for patients with HBV-DNA greater than 500 IU/mL, at least one week of antiviral treatment is required before randomization (only nucleoside analogs such as entecavir, tenofovir disoproxil fumarate, and tenofovir alafenamide tablets are allowed), and the viral copy number should be reduced by more than 10 times compared to before treatment. For HBV infected individuals, antiviral treatment must be received throughout the study period. Patients who are positive for hepatitis C virus (HCV)-RNA must receive antiviral treatment according to the treatment guidelines.
7. Serum bilirubin should be ≤2.0 times the upper limit of normal (ULN); this condition does not apply to patients with confirmed Gilbert's syndrome. Any clinically significant biliary obstruction must be resolved before enrollment in the study.
8. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) should be ≤2.5 times the ULN. For patients with liver metastases, ALT and AST should be ≤5 times the ULN.

Exclusion Criteria:

1. Have an active autoimmune disease or a history of autoimmune disease that may recur (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism).
2. Use of immunosuppressants or systemic corticosteroid therapy for the purpose of immunosuppression within 2 weeks prior to treatment (dose >10mg/day prednisone or other equivalent efficacy corticosteroids).
3. Patients with congenital or acquired immune function deficiency (such as HIV-infected individuals).
4. Have a history of other primary malignant tumors, except for the following situations: malignant tumors treated with curative intent, known to be inactive for ≥5 years prior to the first study intervention and with a low potential risk of recurrence; basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or malignant melanoma in situ that has been treated with potentially curative intent; or in situ cancer that has been adequately treated with no evidence of disease.
5. Known allergy to any study drug or excipients.
6. Participation in other drug clinical studies within the past 4 weeks.
7. Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (mRecist）(ORR) | an average of 1 year
  According to mRECIST to evaluate the proportion of patients with CR and PR in the total number of patients.
Progression-free survival | an average of 1 year
  Patients' progression-free survival after switching to the new treatment regimen is the time between the start of the change and tumor recurrence or death, whichever occurs first

SECONDARY OUTCOMES:
Disease control rate (DCR) | an average of 1 year
  Disease control rate (DCR)
Overall Survival (OS) | an average of 1.5 year
  The time from the date of initiation of the drug donafenib until the date of death from any cause
Incidence of adverse events and serious adverse events | an average of 1.5 year
  Incidence of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Huang, Principal Investigator — Tongji Hospital

IPD SHARING:
Plan to Share IPD: No